CLINICAL TRIAL: NCT05684965
Title: A First-in-Human, Multicenter, Phase 1/2, Open-Label Study of XTX301 in Patients With Advanced Solid Tumors
Brief Title: XTX301 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xilio Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XTX301-01/02-001
Record Dates: First submitted 2022-12-21; First posted 2023-01-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 - XTX301 Monotherapy Dose Escalation and Pharmacodynamics Expansion (Experimental): Part 1A Dose Escalation of XTX301 administered in ascending doses to patients with advanced solid tumors to assess the safety and tolerability and determine/define MTD and/or the highest recommended Phase 2 dose (RP2D).
  Part 1B Evaluation of XTX301 in patients with selected advanced solid tumors to further characterize the pharmacodynamics profile of XTX301.
  Interventions: Drug: XTX301
- Phase 2 - XTX301 Monotherapy Dose Expansion in Disease-Specific Cohorts (Experimental): Phase 2 will further evaluate the safety and antitumor activity/efficacy of XTX301 monotherapy in disease-specific expansion cohorts of patients with select tumors, namely:
  * Cohort 2A: head and neck squamous cell carcinoma (HNSCC)
  * Cohort 2B: melanoma (patients with uveal melanoma are excluded)
  * Cohort 2C: non-small cell lung cancer (NSCLC)
  * Cohort 2D: ovarian cancer
  * Cohort 2E: castrate-resistant prostate cancer (CRPC)
  * Cohort 2F: triple-negative breast cancer (TNBC)
  Interventions: Drug: XTX301

INTERVENTIONS:
Drug: XTX301 — XTX301 monotherapy

SUMMARY:
This is a first-in-human, multicenter, Phase 1/2, open-label study designed to evaluate the safety and tolerability of XTX301 as monotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, multicenter, Phase 1/2, open-label study designed to evaluate the safety, tolerability, PK, PD, immunogenicity, and antitumor activity/efficacy of XTX301, a tumor-activated interleukin-12, as monotherapy in patients with advanced solid tumors.

Phase 1. Part 1A will examine XTX301 monotherapy in a standard 3+3 dose escalation design. Based on the results of Part 1A, patients with select advanced solid tumors will be enrolled in Part 1B, which will evaluate XTX301 monotherapy in relation to specific PD biomarkers.

Phase 2 will further evaluate the safety and antitumor activity/efficacy of XTX301 monotherapy in disease-specific expansion cohorts of patients with select tumors, namely: head and neck squamous cell carcinoma (HNSCC), melanoma (patients with uveal melanoma are excluded), non-small cell lung cancer (NSCLC), ovarian cancer, castrate-resistant prostate cancer (CRPC), triple-negative breast cancer (TNBC)

ELIGIBILITY:
Inclusion Criteria:

• Disease Criteria: Part 1A - Any histologically or cytologically confirmed solid tumor malignancy that is locally advanced or metastatic and has failed standard therapy, standard therapy does not confer survival benefit, or standard therapy is not available.

Part 1B- Any histologically or cytologically confirmed solid tumor malignancy among the tumor types outlined below, that is locally advanced or metastatic and has failed standard therapy, standard therapy does not confer survival benefit, or standard therapy is not available. Patients with the following tumor types are eligible for Part 1B: melanoma, NSCLC, HNSCC, TNBC, cervical cancer, microsatellite instability high/mismatch repair deficient (MSI-H/dMMR) colorectal cancer, or MSI-H/dMMR endometrial cancer. Note: Based on evolving internal and external data, the Sponsor may decide to open a "backfill cohort" in Part 1B for patients with any of the following solid tumors: prostate cancer, ovarian cancer, pancreatic cancer, microsatellite stable colorectal cancer, T-cell lymphoma.

Phase 2 - All patients must have measurable disease at baseline per RECIST 1.1. Additional disease-specific criteria per cohort are as follows:

i. Cohort 2A: head and neck squamous cell carcinoma (HNSCC). Must have histologically or cytologically confirmed locally recurrent or metastatic HNSCC previously treated with 1 to 2 lines of therapy. Unless contraindicated, prior therapy must have included PD-1/PD-L1 inhibitor and/or platinum-based chemotherapy per local and institutional standard of care.

ii. Cohort 2B: melanoma. Must have unresectable or metastatic melanoma previously treated with 1 to 2 lines of therapy in the recurrent or metastatic setting. Unless contraindicated, prior therapy must have included a PD-1/PD-L1 inhibitor alone or in combination. Patients with known BRAF V600-activating mutation must have previously received targeted therapy per local and institutional standard of care. Note: patients with uveal melanoma are excluded.

iii. Cohort 2C: non-small cell lung cancer (NSCLC). Must have histologically confirmed locally advanced or metastatic NSCLC previously treated with 1 to 2 lines of therapy. Unless contraindicated, prior therapy must have included a PD1/PD-L1 inhibitor and a platinum-based regimen, given either concurrently or separately per local and institutional standard of care. Patients with known genomic alteration for which a targeted therapy is approved (e.g. ROS1 fusion, NTRK fusion, BRAF V600E mutation, EGFR mutation, or ALK fusion) must have been previously treated with relevant targeted therapy per local and institutional standard of care.

iv. Cohort 2D: ovarian cancer. Must have histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer with current platinum-resistant disease per investigator's assessment (e.g. patient is not eligible for further platinum-containing treatment). Patients must have previously experienced a response lasting at least 180 days to first-line platinum-based therapy. Patients who have been unable to tolerate platinum therapy are also eligible. Unless contraindicated, patients with known BRCA mutation must have received a poly(ADP-ribose) polymerase (PARP) inhibitor.

v. Cohort 2E: castrate-resistant prostate cancer (CRPC). Must have metastatic CRPC previously treated with an androgen receptor pathway inhibitor (e.g. abiraterone, enzalutamide, darolutamide, or apalutamide) and/or chemotherapy per local and institutional standard of care. Baseline total testosterone must be ≤ 50 ng/dL (≤ 2.0 nM), and surgical or ongoing medical castration must be maintained throughout the duration of the study.

vi. Cohort 2F: triple-negative breast cancer (TNBC). Must have metastatic TNBC with disease relapse after 2 to 4 previous lines of therapy per local and institutional standard of care. Neoadjuvant and/or adjuvant chemotherapy will count as 1 prior line of therapy. Unless contraindicated, patients with known actionable mutations (e.g. BRCA1 or BRCA2) must have received prior therapy with the corresponding targeted agent per local and institutional standard of care

* ECOG performance status of 0-2 for Phase 1
* ECOG performance status of 0 or 1 for Phase 2
* Adequate organ function
* Tumor tissue samples: Part 1B: patients must have lesions amenable to biopsy and be willing and able to provide fresh tumor biopsies before and after initiation of treatment
* Patients with recent major surgery must have adequately recovered with no ongoing complications from the surgery before receiving study drug

Exclusion Criteria:

* Prior treatment with IL-12 therapy (any form, e.g. recombinant human, prodrug, intratumoral, etc.)
* Known liver metastasis based on imaging
* Possible area of ongoing necrosis (non-disease-related), such as active ulcer, nonhealing wound, or intercurrent bone fracture
* Active primary central nervous system (CNS) malignancy, CNS metastases, and/or carcinomatous meningitis
* Active autoimmune disease
* History of Grade ≥ 3 immune-related adverse events associated with prior immunotherapy unless these were adequately resolved with therapy within 14 days
* A diagnosis of immunodeficiency; receiving chronic systemic therapy exceeding prednisone 10 mg daily or equivalent or any other form of immunosuppressive therapy within 7 days before the first dose of study drug
* Active hepatitis B or active hepatitis C infection
* Prior treatment with gene therapy, organ transplant, or hematopoietic stem-cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Part 1A only) | From the first dose of the study drug at Cycle 1 Day 1 up to next applicable cycle visit (Cycle 2 Day 1 or Cycle 3 Day 1). Approximately 21 to 42 days. Each cycle is 21 days.
Incidence of treatment-emergent adverse events (TEAEs) and changes in clinical laboratory values | Up to 24 months
Investigator-assessed objective response rate (ORR) per RECIST 1.1 (Phase 2 only) | up to 24 months

SECONDARY OUTCOMES:
Plasma concentrations of XTX301 | Up to 24 months
Maximum observed plasma concentration (Cmax) | Up to 24 months
Time of maximum observed concentration (Tmax) | Up to 24 months
Trough concentration (Ctrough) | Up to 24 months
Area under the curve (AUC) | Up to 24 months
Half-life (T1/2) | Up to 24 months
Systemic clearance (CL) | Up to 24 months
Volume of distribution (Vd) | Up to 24 months
Antidrug antibody (ADA) occurrence and titer in serum | Up to 24 months
Investigator-assessed objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase 1 only) | Up to 24 months
Duration of response (DOR) (Phase 2 only) | up to 24 months
Disease control rate (Phase 2 only) | up to 24 months
Progression-free survival (PFS) (Phase 2 only) | up to 24 months
Overall survival (OS) (Phase 2 only) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Yale Cancer Center, New Haven, Connecticut
  - HealthPartners Frauenshuh Cancer center, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Gabrail Pharmacology Phase 1 Research Center, Canton, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center-Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tranquil Clinical Research, Webster, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No